CLINICAL TRIAL: NCT01339052
Title: A Phase II Study of BKM 120 for Patients With Recurrent Glioblastoma and Activated PI3K Pathway
Brief Title: Phase II Study of BKM120 for Subjects With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Y. Wen, MD (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Novartis Pharmaceuticals (Industry); M.D. Anderson Cancer Center (Other); Memorial Sloan Kettering Cancer Center (Other); University of California, San Francisco (Other); University of California, Los Angeles (Other); University of Utah (Other)
Responsible Party: Sponsor-Investigator, Patrick Y. Wen, MD, Director, Center For Neuro-Oncology, Dana-Farber/Brigham and Women's Cancer Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-033; CBKM120XUS07T (Other: Novartis)
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Glioblastoma
Keywords: BKM120; Brain tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — NVP-BKM120; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Surgical subjects (Experimental): Subjects scheduled for surgery
  BKM120: 100 mg once daily, orally, for 8-12 days prior to surgery
  Surgery: Surgery
  BKM120: 100 mg once daily, orally, for 28-day cycles
  Patients continued treatment until disease progression or unacceptable toxicity.
  Interventions: Drug: BKM120; Procedure: Surgery
- Cohort 2: Non-surgical subjects (Experimental): Subjects not candidates for surgery
  BKM120: 100 mg once daily, orally, for 28-day cycles
  Patients continued treatment until disease progression or unacceptable toxicity.
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120
  Other Names: Busparlisib
Procedure: Surgery — Surgery
  Arms: Cohort 1: Surgical subjects

SUMMARY:
BKM120 is a newly discovered drug that has been used in other research studies. Information from those other research studies suggests that BKM120 may help to slow or stop the growth of malignant gliomas. The purpose of this study is to see how well BKM120 works in patients with malignant gliomas. Patients on this study will be treated in two groups: patients who are going to receive surgery and those who will not receive surgery. This study is trying to determine how effective BKM120 is in stopping cancer cells from growing. For patients receiving surgery the research will also try to determine if an effective level of BKM120 can penetrate the brain before surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Cohort 1

Primary Objectives

* Evaluate PI3K pathway modulation due to BKM120 in tumor tissue
* Evaluate BKM120 concentration in tumor tissue, plasma, and cerebrospinal fluid

Secondary Objectives

* Evaluate effects of BKM120 on tumor cell proliferation and tumor cell death
* Investigate the safety profile of BKM120 in this population
* Investigate pharmacokinetics of BKM120 in this population

Exploratory Objectives

* Correlate FDG-PET and FLT-PET with pharmacodynamic effects and 6-month progressive-free survival (PFS6)
* Determine the effects of BKM120 on primary GBM cell lines derived from participants and correlate with participant benefit from BKM120 treatment

Cohort 2

Primary Objective

* Investigate the treatment efficacy as measured by 6-month progressive-free survival (PFS6)

Secondary Objectives

* Investigate the radiographic response, progression free survival, overall survival
* Investigate the safety profile efficacy of BKM120 in this population

Exploratory Objectives

* Correlate benefit from BKM120 treatment with molecular genotype of tumor (using immunohistochemistry, mutation analysis and RNA expression profiling), and whole blood proteomics
* Correlate benefit from BKM120 treatment with circulating angiogenic biomarkers
* Utilize advance MRI (perfusion, permeability, diffusion imaging) to determine the effects of BKM120 on tumor vasculature and to correlate with benefit from BKM120 treatment

STATISTICAL DESIGN:

Cohort 1

The primary endpoint for Cohort 1 is modulation of PI3 kinase pathway based on change in immunohistochemistry (IHC) scoring for pAKT. Modulation in scoring as measured by reduction of staining intensity score of one degree or more was reported as a positive response to drug. This portion of the trial would be considered a success if 9 or more participants of 15 participants showed a response. There was a 94% chance of this occurring if the true response rate was 75% and only a 10% chance of this occurring if the true response rate was 40%.

Cohort 2

The primary endpoint for Cohort 2 is the proportion of participants progression free at 6 months (PFS6). Historical comparison data suggest that ineffective therapies in recurrent GBM have a PFS6 rate of approximately 9-16% (Wong 1999; Lamborn 2008). This trial was sized to differentiate between a 15% versus a 32% PFS6. With a total sample size of 50 participants, this design yields at least 90% power with a one sided alpha < 0.1 to detect a true PFS6 rate of at least 32%. If the number of successes was ≥ 12, the therapy would be considered worthy of further study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to understand and be willing to sign a written informed consent document.
* Subjects must be able to adhere to the dosing and visit schedules, and agree to record medication times accurately and consistently in a daily diary.
* Participants must be at least 18 years old.
* Participants must have a Karnofsky performance status (KPS) ≥ 60. Nature of illness and treatment history
* Participants must have histologically confirmed glioblastoma or variants. Participants will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of glioblastoma or variants is made.
* Participants may have had treatment for no more than 1 prior relapse(NOTE: Relapse is defined as progression following initial therapy (i.e., radiation ± chemotherapy)). The intent therefore is that patients had no more than 2 prior therapies (initial and treatment for 1 relapse). If the participant had a surgical resection for relapsed disease and no antitumor therapy was instituted for up to 12 weeks, and the participant undergoes another surgical resection, this is considered as a second relapse. For participants who had prior therapy for a low-grade glioma, the surgical diagnosis of a high-grade glioma will be considered the first relapse).
* Participants must have shown unequivocal evidence for tumor progression by MRI or CT scan.
* For Cohort 2, CT or MRI within 14 days prior to start of study drug. MRIs should include vascular imaging when possible. For Cohort 2, corticosteroid dose must be stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the screening MRI or CT scan and the start of treatment, a new baseline MRI or CT is required. For Cohort 1 subjects, CT or MRI should be performed ideally within 14 days prior to study registration, but because the screening MRI for this subset of subjects will not be used for evaluation of response, it is acceptable for this MRI/CT to have been performed greater than 14 days prior to registration if unavoidable. Furthermore, for this same reason, fluctuation in corticosteroid dose around this MRI does not warrant repeat scan so long as there is documented unequivocal evidence of tumor progression available.
* For Cohort 2, Immunohistochemical or genetic analysis on tumor tissue from a prior surgery must demonstrate activation of the PI3K pathway through one of the following: PIK3CA mutation of PIK3R1 mutation, PTEN negativity (<10% of tumor cells staining) oh immunohistochemistry, PTEN mutation (any), homozygous deletion of PTEN
* Participants must have failed prior radiation therapy and must have an interval of at least 12 weeks from the completion of radiation therapy to study entry.
* Participants must have recovered to a grade 0 or 1 from the toxic effects of prior therapy (with the exception of lymphopenia which is common after therapy with temozolomide).
* From the projected start of scheduled study treatment, the following time periods must have elapsed: 4 weeks or 5 half-lives (whichever is shorter)from any investigational agent, 4 weeks from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies, or 4 weeks or 5 half-lives (whichever is shorter) from other anti-tumor therapies.
* Participants with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of progressive disease based upon nuclear imaging, MR spectroscopy, perfusion imaging or histopathology.
* Participants having undergone recent resection of recurrent or progressive tumor will be eligible for Cohort 2 as long as the following conditions apply: a) They have recovered from the effects of surgery; b) Residual disease following resection of recurrent tumor is not mandated for eligibility. To best assess the extent of residual disease postoperatively, an MRI or CT scan should ideally been performed no later than 96 hours following surgery or at least 28-days postoperatively, but scans performed outside of this window are considered acceptable if no alternative is available. In either case, the baseline/screening MRI must be performed within 14 days prior to registration. If the participant is taking corticosteroids, the dose must be stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the screening MRI or CT scan and the start of treatment, a new baseline MRI or CT is required.
* Participants must have sufficient tissue from prior surgery for confirmation of diagnosis and correlative studies. Submission of tissue is to occur within 30 days after registration. The following amount of tissue is required: a) 25 unstained formalin fixed paraffin embedded (FFPE) sections (standard 4-5 micrometer thickness AND b)one of the following: i) At least 200 micrograms of frozen tissue OR ii)At least 10 (preferably 20) unstained FFPE sections of 10 micrometer thickness OR iii) At least 8 tissue cores from an FFPE block (200 micrometer total thickness of tissue from a block with a total surface area of 0.5 cm2)
* Clinical laboratory tests within 14 days prior to enrollment meeting the criteria listed in the protocol
* Cardiovascular assessment: baseline MUGA or Echocardiogram must demonstrate LVEF ≥ 50 %
* Electrocardiogram must demonstrate QTc interval of less than 480 msec
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective contraception (defined in protocol) during study treatment and for 16 weeks after study discontinuation.
* Women of child-bearing potential must have a negative serum pregnancy test at screening and within 48 hours prior to dosing with the study drug.
* Fertile males, defined as all males physiologically capable of conceiving offspring, must use condom during study treatment and for 16 weeks after study discontinuation and should not father a child in this period.
* Female partner of male study subject should use highly effective contraception while receiving study agent and for 16 weeks after final dose of study therapy.

Cohort 1 Inclusion Criteria (In addition to the general eligibility criteria, participants in the Cohort 1 preoperative portion of the study must meet the following criteria on screening examination to be eligible):

* A participant who is deemed by the site Investigator to be an appropriate candidate for surgical resection may be enrolled in the Cohort 1 preoperative study.
* There must be sufficient recurrent tumor to allow at least 400mg of tissue to be collected ( 2 X 0.5 cm3) for pharmacokinetic and pharmacodynamic analysis.
* Central Immunohistochemical analysis (by Dr. Ligon at DFCI) on tumor tissue from an earlier surgery must indicate pAKT positivity (1-2+ on a 0-2+ scale). [Cohort I patients' tissue may also demonstrate activation of the PI3K pathway via one of the criteria listed for Cohort 2 participants, but this is not mandatory.]

Exclusion Criteria:

* Participants who have received prior treatment with a P13K inhibitor, AKT inhibitor, mTOR inhibitor (e.g. rapamycin, MK2206, perifosine etc.).
* Participants who have received anti-angiogenic or anti-VEGF targeted agents (e.g. bevacizumab, cediranib, aflibercept, vandetanib, XL184, sunitinib etc).
* Participants taking an enzyme-inducing anti-epileptic drug (EIAED): phenobarbital, phenytoin, fosphenytoin, primidone, carbamazepine, oxcarbazepine, eslicarbazepine, rufinamide, and felbamate. Participant must be off any EIAEDs for at least two weeks prior to starting study drug. A list of EIAED and other inducers of CYP3A4 is provided in Table C-3 of Appendix C of the protocol.
* Participants taking a drug known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A (protoocol Appendix C). Participant must be off CYP3A inhibitors and inducers for at least two weeks prior to starting study drug. NOTE: participants must avoid consumption of Seville orange (and juice), grapefruit or grapefruit juice, grapefruit hybrids, pummelos and exotic citrus fruits from 7 days prior to the first dose of study drug and during the entire study treatment period due to potential CYP3A4 interaction.
* Requirement of more than 8mg of dexamethasone daily.
* Participants taking drugs with known risk to promote QT prolongation and Torsades de Pointes (refer to protocol).
* Participants receiving any other investigational agents.
* Current use of herbal preparations/medications, including but not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, ginseng. Participants should stop using these herbal medications 7 days prior to first dose of study drug.
* Current use of warfarin sodium or any other coumadin-derivative anticoagulant. Participant must be off Coumadin-derivative anticoagulants for at least 7 days prior to starting study drug. Low molecular weight heparin is allowed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BKM120.
* History of intratumoral or peritumoral hemorrhage if deemed significant by the treating physician.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, chronic liver disease (e.g., cirrhosis, hepatitis), chronic renal disease, pancreatitis, chronic pulmonary disease, or psychiatric illness/social situations that would limit compliance with study requirements. Subjects must be free of any clinically relevant disease (other than glioma) that would, in the Investigator's opinion, interfere with the conduct of the study or study evaluations.
* Individuals with a history of a different malignancy except for the following circumstances: if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy, individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Known diagnosis of human immunodeficiency virus (HIV) infection
* Participants with history of protocol specified mood disorders as judged by the Investigator or a psychiatrist, or as result of participant's screening mood assessment questionnaire
* Participants with diarrhea ≥ CTCAE grade 2
* Participant has active cardiac disease including any of the following: Angina pectoris that requires the use of anti-anginal medications; Ventricular arrhythmias except for benign premature ventricular contractions; Supraventricular and nodal arrythmias requiring a pacemaker or not controlled with medication; Conduction abnormality requiring a pacemaker; Valvular disease with document compromise in cardiac function; Symptomatic pericarditis
* Participant has a history of cardiac dysfunction including any of the following: Myocardial infraction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function; History of documented congestive heart failure (New York Heart Association functional classification III-IV; c)Documented cardiomyopathy; d) Congenital long QT syndrome
* Participants with poorly controlled diabetes mellitus (glycosylated hemoglobin > 8%) or poorly controlled steroid-induced diabetes mellitus (glycosylated hemoglobin > 8%)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or extensive small bowel resection). Participants with unresolved diarrhea will be excluded as previously indicated.
* Participants who have undergone major systemic surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - UT, MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wen PY, Touat M, Alexander BM, Mellinghoff IK, Ramkissoon S, McCluskey CS, Pelton K, Haidar S, Basu SS, Gaffey SC, Brown LE, Martinez-Ledesma JE, Wu S, Kim J, Wei W, Park MA, Huse JT, Kuhn JG, Rinne ML, Colman H, Agar NYR, Omuro AM, DeAngelis LM, Gilbert MR, de Groot JF, Cloughesy TF, Chi AS, Roberts TM, Zhao JJ, Lee EQ, Nayak L, Heath JR, Horky LL, Batchelor TT, Beroukhim R, Chang SM, Ligon AH, Dunn IF, Koul D, Young GS, Prados MD, Reardon DA, Yung WKA, Ligon KL. Buparlisib in Patients With Recurrent Glioblastoma Harboring Phosphatidylinositol 3-Kinase Pathway Activation: An Open-Label, Multicenter, Multi-Arm, Phase II Trial. J Clin Oncol. 2019 Mar 20;37(9):741-750. doi: 10.1200/JCO.18.01207. Epub 2019 Feb 4. PMID 30715997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from September 2011 through February 2014.
Groups:
- Cohort 1: Surgical Subjects: Subjects scheduled for surgery
  BKM120: 100 mg once daily, orally, for 8-12 days prior to surgery
  Surgery: Surgery
  BKM120: 100 mg once daily, orally, for 28-day cycles
  Participants continued treatment until disease progression or unacceptable toxicity.
- Cohort 2: Non-surgical Subjects: Subjects not candidates for surgery
  BKM120: 100 mg once daily, orally, for 28-day cycles
  Participants continued treatment until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort 1: Surgical Subjects | Cohort 2: Non-surgical Subjects
Started | 15 | 50
Measurable Disease (Measurable disease post-surgery for Cohort 1 participants.) | 11 | 40 (Radiographic response evaluated on participants with measurable disease only.)
Evaluable Tumor Sample at Surgery | 14 | 0 (Milestone is not relevant for non-surgical cohort.)
Evaluable Plasma Sample at Surgery | 13 | 0 (Milestone is not relevant for non-surgical cohort.)
Completed (Since treatment was not of fixed duration, all participants were considered as 'Not Completed'.) | 0 | 0
Not Completed | 15 | 50
Not completed — Disease progression | 13 | 46
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Surgical Subjects | Cohort 2: Non-surgical Subjects | Total
Number analyzed (Participants) | 15 | 50 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 43 | 56
  >=65 years | 2 | 7 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 13 | 17
  Male | 11 | 37 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 11 | 35 | 46
  Unknown or Not Reported | 4 | 13 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 32 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 15 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 50 | 65
Karnofsky performance status (KPS) [Count of Participants; unit: Participants] — 'Karnofsky Performance Status' (KPS) scale: 100 = Normal; no complaints; no evidence of disease; 90 = Able to carry on normal activity; minor signs or symptoms of disease; 80 = Normal activity with effort; some sign or symptoms of disease; 70 = Cares for self; unable to carry on normal activity or do active work.
  Participants
    70 | 1 | 3 | 4
    80 | 2 | 15 | 17
    90 | 10 | 23 | 33
    100 | 2 | 9 | 11
Current Tumor Diagnosis [Count of Participants; unit: Participants]
  Glioblstoma Multiforme (GBM) | 15 | 47 | 62
  Gliosarcoma | 0 | 3 | 3
Initial Tumor Diagnosis [Count of Participants; unit: Participants]
  Glioblastoma Multiforme (GBM) | 13 | 41 | 54
  Anaplastic Astrocytoma (AA) merging w Glioblastoma | 1 | 0 | 1
  Gr4 Right Parietal Glioma | 1 | 0 | 1
  Astrocytoma | 0 | 1 | 1
  Anaplastic Astrocytoma (AA) | 0 | 3 | 3
  Gemistocytic Astrocyoma | 0 | 1 | 1
  Glioma consistent w/ mixed Oligoastrocytoma | 0 | 1 | 1
  Gliosarcoma | 0 | 1 | 1
  High grade astrocytoma/glioblastoma | 0 | 1 | 1
  Oligodendroglioma | 0 | 1 | 1
PTEN Status at Registration via Central Path Review [Count of Participants; unit: Participants]
  PTEN Negative | 7 | 34 | 41
  Not PTEN Negative | 8 | 12 | 20
  PTEN loss by FISH | 0 | 1 | 1
  PTEN Mutant | 0 | 1 | 1
  Unknown/Pending | 0 | 2 | 2
pAKT StatusStatus at Registration via Central Path Review [Count of Participants; unit: Participants]
  pAKT Positive | 15 | 39 | 54
  pAKT Negative | 0 | 2 | 2
  Unknown/Pending | 0 | 9 | 9
Mutation Status at Registration [Count of Participants; unit: Participants]
  PIK3CA mutation | 1 | 2 | 3
  Negative | 0 | 1 | 1
  Unknown/Pending | 14 | 47 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in pAKT (S473) Immunohistochemistry (IHC) Score From Baseline to Surgery [Cohort 1]
Description: pAKT response was determined by pathologist-performed semi-quantitative IHC scoring for pAKT using previously established methods for glioblastoma (GBM) patients. Sample staining scored for intensity on a 0-2+ scale (0 none, 1+ weak positive, 2+ strong positive). Change in pAKT IHC score was the difference in score from baseline to surgery. Participants were classified into 3 groups: a reduction of staining score of one degree or more (considered a response), an increase in score and no change in score.
Time Frame: Samples were collected at baseline and at surgery (resected surgical tumor specimen) which occurred after up to 12 days of BKM120 treatment.
Population: The analysis dataset is comprised of all treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Surgical Subjects
Number analyzed (Participants) | 15
Participants
  reduced pAKT (S473) IHC Score | 6
  increased pAKT (S473) IHC Score | 1
  no change in pAKT (S473) IHC Score | 7
  Unevaluable | 1

2. Primary Outcome: 6-Month Progression-Free Survival (PFS6) [Cohort 2]
Description: PFS6 is the proportion of participants remaining alive and progression-free at 6-months from cycle 1 day 1 of BKM120 treatment. Progressive disease is defined using RANO (Response Assessment in Neuro-Oncology) criteria (Wen et al JCO 2010), which takes modified Macdonald Criteria and adds assessment of non-enhancing lesions. Per RANO, progressive disease (PD) is defined either as > 25% increase in sum of the products of perpendicular diameters of enhancing lesions on stable or increasing doses of corticosteroids, or one or more of the of the following: 1) Significant increase in T2/FLAIR non-enhancing lesion on stable or increasing doses of corticosteroids steroids not due to co-morbid events; 2) Any new lesion; 3) Clear clinical deterioration not attributable to other causes apart from the tumor; or 4) Failure to return for evaluation due to death or deteriorating condition.
Time Frame: Participants were assessed radiologically every other cycle on treatment; Relevant for this outcome is up to month 6 evaluation.
Population: The analysis dataset is comprised of all treated participants.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2: Non-surgical Subjects
Number analyzed (Participants) | 50
proportion of participants | 0.08 [0.028 to 0.174]

3. Primary Outcome: BKM120 Brain-to-Plasma Ratio at Time of Surgery [Cohort 1]
Description: Levels of BKM120 were determined by liquid chromatography coupled with tandem mass spectrometry. BKM120 tumor-to-plasma ratio at time of surgery was calculated based on these levels.
Time Frame: Samples were collected at surgery (surgical tumor specimen and plasma sample) which occurred after up to 12 days of BKM120 treatment.
Population: The analysis dataset is comprised of participants with a paired plasma and brain tumor sample (evaluable). Participants missing a brain tumor sample (n=1) or plasma sample (n=2) are excluded from the calculation.
Measure: Geometric Mean (Full Range); unit: ratio tumor-to-plasma
Arm/Group | Cohort 1: Surgical Subjects
Number analyzed (Participants) | 13
ratio tumor-to-plasma | 1.00 [0.18 to 8.44]

4. Primary Outcome: BKM120 Tumor Tissue Concentration at Time of Surgery [Cohort 1]
Description: Levels of BKM120 were determined by liquid chromatography coupled with tandem mass spectrometry.
Time Frame: Samples were collected at surgery (resected surgical tumor specimen) which occurred after up to 12 days of BKM120 treatment.
Population: The analysis dataset is comprised of all participants with a resected surgical tumor specimen (evaluable).
Measure: Geometric Mean (Full Range); unit: ng/gm
Arm/Group | Cohort 1: Surgical Subjects
Number analyzed (Participants) | 14
ng/gm | 590 [86 to 6947]

5. Primary Outcome: BKM120 Plasma Concentration at Time of Surgery [Cohort 1]
Description: Levels of BKM120 were determined by liquid chromatography coupled with tandem mass spectrometry.
Time Frame: Samples were collected at surgery which occurred after up to 12 days of BKM120 treatment.
Population: The analysis dataset is comprised of all participants with a plasma sample at surgery (evaluable).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Surgical Subjects
Number analyzed (Participants) | 13
ng/mL | 585 (192)

6. Secondary Outcome: % Ki-67 Reduction Using Immunohistochemistry (IHC) [Cohort 1]
Description: Tumor cell proliferation and tumor cell death was using immunohistochemistry for Ki-67 based on established methods. Percent reduction was based on Ki-67 levels at baseline and at surgery.
Time Frame: Samples were collected at baseline (archival tumor specimen) and at surgery (surgical tumor specimen) which occurred after up to 12 days of BTK120 treatment.
Population: The analysis dataset is comprised of all participants with a resected surgical tumor specimen (evaluable).
Measure: Median (Full Range); unit: % reduction
Groups:
- Cohort I: Surgical Subjects: Subjects scheduled for surgery
  BKM120: 100 mg once daily, orally, for 8-12 days prior to surgery
  Surgery: Surgery
  BKM120: 100 mg once daily, orally, for 28-day cycles
  Participants continued treatment until disease progression or unacceptable toxicity.
Arm/Group | Cohort I: Surgical Subjects
Number analyzed (Participants) | 14
% reduction | 11 [-81 to 100]

7. Secondary Outcome: Radiographic Response [Cohort 2]
Description: Radiographic response was based on RANO (Response Assessment in Neuro-Oncology) criteria. Per RANO, complete response (CR): 1) Complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks, 2) No new lesions, 3) All lesions assessed using the same techniques as baseline, 4) No steroid use (or on physiologic replacement doses only), 5) Stable or improved non-enhancing (T2/FLAIR) lesions and 6) Stable or improved clinically; partial response (PR): 1) >/= 50% decrease compared to baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions (sum LD) sustained for at least 4 weeks and 2) No progression; progressive disease (PD): 1) > 25% increase sum LD and/or 2) significant increase in T2/FLAIR, 3) any new lesion, 4) clear clinical deterioration; stable disease (SD): none of the above.
Time Frame: Participants were assessed radiologically every other cycle on treatment. Cohort 2 participants were on treatment up to 9.2 months.
Population: Only those participants who had measurable disease present at baseline and received at least one dose of therapy are considered evaluable for radiographic response
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Non-surgical Subjects
Number analyzed (Participants) | 40
Participants
  Stable Disease | 16
  Progressive Disease | 22
  Not Evaluable | 2

8. Secondary Outcome: Maximum Observed Plasma Concentrations (Cmax) of BKM120 Day 1 and Day 8 [Cohort 1]
Description: Plasma concentrations of BKM120 were analyzed by a validated liquid chromatography-tandem mass spectrometry assay developed by Novartis Pharma AG. Standard Pk parameters were determined using non-compartmental methods.
  NOTE: This outcome measure was previously titled: "Investigate Pharmacokinetics of BKM120 in This Population by Comparing Maximum Plasma Concentrations (Cmax) From Day 1 to Day 8"
Time Frame: On days 1 and 8 (+/- 1 day) prior to surgery, 5 blood samples were collected at the following timepoints: pre-dose, and at 0.5, 1.5, 3, and 5 hours post-dose.
Population: The analysis dataset is comprised of all treated patients.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Surgical Subjects
Number analyzed (Participants) | 15
ng/mL
  Day 1 | 471 (147)
  Day 8 | 820 (192)

9. Secondary Outcome: Cmax Accumulation Ratio of BKM120 Day 1 and Day 8 Ratio [Cohort 1]
Description: Plasma concentrations of BKM120 were analyzed by a validated liquid chromatography-tandem mass spectrometry assay developed by Novartis Pharma AG. Standard Pk parameters were determined using non-compartmental methods. The accumulation ratio is day 8/day 1.
Time Frame: as for outcome 8
Population: The analysis dataset is comprised of all treated patients.
Measure: Mean (Full Range); unit: ratio day 8/day 1
Arm/Group | Cohort I: Surgical Subjects
Number analyzed (Participants) | 15
ratio day 8/day 1 | 1.88 [1.377 to 2.383]

10. Secondary Outcome: Area Under the Concentration Curve From Time 0 to Last Concentration (AUC0-5h) of BKM120 Day 1 and Day 8 [Cohort 1]
Description: Plasma concentrations of BKM120 were analyzed by a validated liquid chromatography-tandem mass spectrometry assay developed by Novartis Pharma AG. Standard Pk parameters were determined using non-compartmental methods.
  NOTE: This outcome measure was previously titled: "Investigate Pharmacokinetics of BKM120 in This Population by Comparing the Drug Exposure Area Under the Curve (AUC0-5h) From Day 1 to Day 8"
Time Frame: as for outcome 8
Population: The analysis dataset is comprised of all treated patients.
Measure: Mean (Standard Deviation); unit: ug*h/mL
Arm/Group | Cohort 1: Surgical Subjects
Number analyzed (Participants) | 15
ug*h/mL
  Day 1 | 1.42 (0.50)
  Day 8 | 3.27 (1.43)

11. Secondary Outcome: AUC0-5h Accumulation Ratio of BKM120 Day 1 and Day 8 [Cohort 1]
Description: as for outcome 9
Time Frame: as for outcome 8
Population: The analysis dataset is comprised of all treated patients.
Measure: Mean (Full Range); unit: ratio day 8/day 1
Arm/Group | Cohort I: Surgical Subjects
Number analyzed (Participants) | 15
ratio day 8/day 1 | 2.42 [1.694 to 3.146]

12. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of BKM120 Day 1 and Day 8 [Cohort 1]
Description: Plasma concentrations of BKM120 were analyzed by a validated liquid chromatography-tandem mass spectrometry assay developed by Novartis Pharma AG. Standard Pk parameters were determined using non-compartmental methods.
Time Frame: as for outcome 8
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Surgical Subjects
Number analyzed (Participants) | 15
hours
  Day 1 | 1.5 [1.5 to 5]
  Day 8 | 1.5 [0.5 to 9]

13. Secondary Outcome: Overall Survival (OS) [Cohort 2]
Description: Overall survival is defined as the time from date of first dose to death or date last known alive and estimated using Kaplan-Meier (KM) methods.
Time Frame: Participants were followed long-term for survival via medical record review. Cohort 2 participants were followed for survival up to 52 months in this study cohort.
Population: The analysis dataset is comprised of all treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2: Non-surgical Subjects
Number analyzed (Participants) | 50
months | 9.8 [8.4 to 12.4]

14. Secondary Outcome: Progression-Free Survival (PFS) [Cohort 2]
Description: PFS is defined as the time from first dose to the earliest documentation of disease progression or death. Participants alive without evidence of PD were censored at the date of last disease assessment. Progressive disease was established based on Response Assessment in Neuro-Oncology (RANO) criteria (Wen et al JCO 2010). See outcome measure #2.
Time Frame: Participants were assessed radiologically every other cycle on treatment and off-treatment via medical record review until death. Cohort 2 participants were followed for progression-free survival up to 12 months in this study cohort.
Population: The analysis dataset is comprised of all treated participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2: Non-surgical Subjects
Number analyzed (Participants) | 50
months | 1.7 [1.4 to 2.7]

15. Secondary Outcome: Grade 3-5 Treatment-Related Toxicity Rate
Description: The percentage of patients who experienced any grade 3-5 treatment-related adverse event based on CTCAEv4 as reported on case report forms.
Time Frame: Adverse events experienced by participants are collected and reported throughout treatment with study drug (from initiation of study medication until 30 days after the last dose of BKM120), maximum timeframe was 2 years.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of patients
Groups:
- Cohorts 1: Surgical Subjects: Subjects scheduled for surgery
  BKM120: 100 mg once daily, orally, for 8-12 days prior to surgery
  Surgery: Surgery
  BKM120: 100 mg once daily, orally, for 28-day cycles
  Patients continued treatment until disease progression or unacceptable toxicity.
- Cohorts 2: Non-surgical Subjects: Subjects not candidates for surgery
  BKM120: 100 mg once daily, orally, for 28-day cycles
  Patients continued treatment until disease progression or unacceptable toxicity.
Arm/Group | Cohorts 1: Surgical Subjects | Cohorts 2: Non-surgical Subjects
Number analyzed (Participants) | 15 | 50
percentage of patients | 40.0 [19.1 to 64.0] | 32.0 [21.2 to 44.5]

ADVERSE EVENTS:
Time Frame: Adverse events experienced by participants are collected and reported throughout treatment with study drug (from initiation of study medication until 30 days after the last dose of BKM120), maximum timeframe was 2 years.
Description: The following are considered 'serious' adverse events (SAEs) per protocol:
  * ALL Grade 5 (fatal) Events
  * ALL Grade 4 (life threatening or disabling) Events - Unless both Expected AND specifically listed in protocol as not requiring reporting
  * ANY Grade 2 (moderate) or Grade 3 (severe) Event that is both Unexpected and deemed at least Possibly Related to study intervention Other AEs: Remaining AEs (maximum grade by toxicity type) without regard to treatment attribution.
Arm/Group | Cohorts 1: Surgical Subjects | Cohorts 2: Non-surgical Subjects
All-Cause Mortality (participants affected / at risk) | 0/15 | 2/50
Serious Adverse Events (participants affected / at risk) | 5/15 | 12/50
Other Adverse Events (participants affected / at risk) | 15/15 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts 1: Surgical Subjects (N=15) | Cohorts 2: Non-surgical Subjects (N=50)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 1 (1)
Lipase Increased (Investigations) | 0 (0) | 3 (3)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 1 (2) | 2 (3)
Weight loss (Investigations) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (2) | 0 (0)
Spasticity (Nervous system disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts 1: Surgical Subjects (N=15) | Cohorts 2: Non-surgical Subjects (N=50)
Hearing Impaired (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (4) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 5 (8) | 12 (15)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 6 (6)
Nausea (Gastrointestinal disorders) | 6 (6) | 8 (8)
Fatigue (General disorders) | 11 (23) | 28 (41)
Irritability (General disorders) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2) | 7 (15)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (9)
Lipase increased (Investigations) | 2 (2) | 8 (9)
Lymphocyte count decreased (Investigations) | 2 (5) | 2 (2)
Platelet count decreased (Investigations) | 3 (4) | 7 (15)
Serum amylase increased (Investigations) | 3 (3) | 5 (8)
White blood cell decreased (Investigations) | 2 (2) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (9) | 25 (66)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (7) | 2 (3)
Agitation (Psychiatric disorders) | 1 (1) | 6 (6)
Anxiety (Psychiatric disorders) | 3 (6) | 11 (18)
Depression (Psychiatric disorders) | 6 (9) | 11 (20)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (9) | 5 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (6)
Hypertension (Vascular disorders) | 0 (0) | 7 (15)
Thromboembolic event (Vascular disorders) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Rash, unspecified (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin/subcutaneous tissue disorders; Other, specify: Significant confluent erythema covering essentia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4)
Chills (General disorders) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 1 (6) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 4 (5)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Eye disorders - Other, specify: Left visual field cut/difficulty (Eye disorders) | 1 (1) | 1 (1)
Eye disorders - Other, specify: Eye Disorder:Dyplopia-Double Vision (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify: Quadranopsia, right (Eye disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Infections and infestations - Other, specify: varicella-zoster virus infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 1 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (7)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 3 (4) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 7 (7)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Dysphasia (Nervous system disorders) | 2 (2) | 9 (10)
Headache (Nervous system disorders) | 2 (2) | 17 (21)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 9 (10)
Nervous system disorders - Other, specify: left tongue deviation (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 4 (6) | 11 (14)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (2) | 6 (6)
Insomnia (Psychiatric disorders) | 1 (1) | 5 (7)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 5 (7)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: mild pain at incision site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Fungal Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 2 (2)
Optic nerve disorder (Eye disorders) | 0 (0) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gait disturbance (General disorders) | 0 (0) | 9 (10)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Weight gain (Investigations) | 0 (0) | 2 (3)
Concentration impairment (Nervous system disorders) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 2 (3)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 4 (4)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Personality change (Psychiatric disorders) | 0 (0) | 2 (2)
Surgical and medical procedures - Other, specify: Surgery (post-treatment craniotomy) (Surgical and medical procedures) | 0 (0) | 2 (2)
Nervous system disorders - Other, specify: Aphasia (Nervous system disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days